CLINICAL TRIAL: NCT03647085
Title: Data Collection Atrial Fibrillation Exploratory Study
Acronym: CAFE
Status: Terminated | Type: Observational
Why Stopped: Due to COVID-19 and resourcing challenges
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C2106
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: atrial fibrillation; atrial flutter; arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Wearable Cardiac Monitor: Patients diagnosed with, and currently in, persistent atrial fibrillation at the time of enrollment and are scheduled for an ablation or cardioversion.
  Interventions: Device: Wearable cardiac monitor
- Group 2 Wearable Cardiac Monitor: Patients diagnosed with, and currently in, paroxysmal atrial fibrillation at the time of enrollment and are scheduled for an ablation or cardioversion.
  Interventions: Device: Wearable cardiac monitor
- Group 3 Wearable Cardiac Monitor: Patients diagnosed with, and currently in, atrial flutter at the time of enrollment and are scheduled for an ablation or cardioversion.
  Interventions: Device: Wearable cardiac monitor

INTERVENTIONS:
Device: Wearable cardiac monitor — Participants will be fitted with a wearable cardiac monitor placed on the skin that measures physiologic signals.

SUMMARY:
To characterize the impact of Atrial fibrillation (AFib) and Atrial Flutter (AFl) on signals measured using a wearable cardiac monitor prototype device.

To evaluate the relationship of AFib/AFl symptom severity with various physiologic signals measured from the wearable cardiac monitor prototype device.

DETAILED DESCRIPTION:
The is a non-randomized feasibility study that will enroll up to 50 participants with an ongoing episode of AFib/AFl and are referred for a cardiac ablation or electrical cardioversion procedure. A maximum of 20 persistent AFib, 20 paroxysmal AFib, and 20 AFl participants will be enrolled, not to exceed 50 total. There will be up to three data collection visits.

Visit 1 will occur on the same day as enrollment and prior to the cardiac ablation or electrical cardioversion procedure. This allows collection of physiologic signals while the patient is in AFib or AFI.

Visit 2 will occur after the cardiac ablation or electrical cardioversion procedure; no earlier than the day after the cardiac ablation or electrical cardioversion procedure and no more than 4 months after the day of the procedure.

Visit 3 is optional, and may be scheduled upon sponsor's request, which will take place at least 5 months after the previous (second) data collection visit.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to provide written informed consent to participate in the trial
* Age 18 years old or greater
* Willing and able to participate in study visits and the required testing
* Diagnosed with paroxysmal AFib or persistent AFib or AFl and scheduled for a cardiac ablation or electrical cardioversion procedure
* Confirmed AFib/AFl at the time of enrollment

Exclusion Criteria:

* Currently enrolled in another clinical trial that may interfere with the placement of study system or include the usage of unapproved drugs
* Participant is pregnant or planning to become pregnant during the study
* Diagnosed with permanent AFib
* Active Implantable Medical Device, e.g. cardiac implantable electronic devices, bladder stimulators, diaphragm stimulators, implantable neuro stimulator, implantable active monitoring devices, implantable active drug administration devices, etc.
* Known allergy to materials used in the study (adhesive tape, ECG electrodes)
* Have a prosthetic cardiac valve or previously underwent cardiac valve surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with paroxysmal AFib or persistent AFib or AFl and scheduled for a cardiac ablation or electrical cardioversion procedure.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Physiologic Signal Detection | 12 months
  Characterize the impact of Atrial fibrillation (AFib) and Atrial Flutter (AFl) on signals measured using a wearable cardiac monitor prototype device.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Johnson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Foundation, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No